CLINICAL TRIAL: NCT04037631
Title: Prospective Clinical Study to Compare Visual Performance Obtained With a New Diagnostic Device
Brief Title: Compare Visual Outcomes Using a New Diagnostic Device
Status: Terminated | Type: Observational
Why Stopped: recruitment
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AT-LISA-tri 839MP BER-401-17
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients without clinically significant age-related cataract
  Interventions: Diagnostic Test: Diagnostic device

INTERVENTIONS:
Diagnostic Test: Diagnostic device — Diagnostic test

SUMMARY:
Evaluation of preoperative corrected distance visual acuity (CDVA) obtained with VirtIOL device compared to postoperative CDVA.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent
* Patients of any gender, aged 18 years to open age
* Assured follow-up examinations
* Healthy eyes without clinically significant age-related cataract

  -Exclusion Criteria:
* Patients unable to meet the limitations of the protocol or likely of non-cooperation during the trial
* Patients whose freedom is impaired by administrative or legal order
* Concurrent participation in another drug or device investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without clinically significant age-related cataract
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity (CDVA) | 3 months after surgery
  Evaluation of CDVA obtained with diagnostic device

CONTACTS AND LOCATIONS:
Locations (1):
- Internationale Innovative Ophthalmologie, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schallhorn SC, Fernandez J, Kaymak H, Gerlach M, Kirchner FO. Prediction of visual outcomes using virtual implantation of a trifocal intraocular lens in presbyopic lens exchange patients. J Cataract Refract Surg. 2025 Feb 1;51(2):133-140. doi: 10.1097/j.jcrs.0000000000001576. PMID 39453845